CLINICAL TRIAL: NCT04370457
Title: Randomized Clinical Trial of the MyPal ePRO-based Early Palliative Care System in Adult Patients With Hematologic Malignancies
Brief Title: MyPal ePRO-based Early Palliative Care System in Adult Patients With Hematologic Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Research and Technology Hellas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MyPAL4Adults
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Chronic Lymphocytic Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Administration of the MyPal ePRO system
  Interventions: Other: Administration of the MyPal ePRO system
- Standard care arm (No Intervention): No further intervention besides standard palliative care approach if needed

INTERVENTIONS:
Other: Administration of the MyPal ePRO system — Patients will be asked to complete self-report questionnaires at baseline, and every month for the first six months and at 12-month follow-up
  Arms: Experimental arm

SUMMARY:
Randomized unblinded interventional clinical trial:

Arm Intervention Experimental arm (n=150): Intervention group Administration of the MyPal ePRO system the intervention group will use the ePRO tools provided in the project.

Standard care arm (n=150): no intervention besides general palliative care if required general palliative care if required.

Patients will be randomly assigned in a 1:1 fashion to use the MyPal system and receive related-intervention versus general palliative care, stratified by cancer type (i.e. CLL vs MDS), using a computer-generated number sequence, which will be concealed until after group assignment.

DETAILED DESCRIPTION:
The MyPal eHealth system coincides with the MyPal intervention. The system will be used primarily by the patients that participate in the intervention arm of the trial and secondarily by the participating healthcare professionals (HCP). Patients participating in the standard arm of the trial won't use the system. Access to the MyPal eHealth system will be granted to the patients and HCP right after their enrollment in the trial. Patients will have access to the system continuously for 12 months; HCP will have access to the system until the end of the trial.

The main modules (software and hardware) of the system are outlined below:

* MyPal smartphone application (app). This is the interface of the patient to the system. The MyPal smartphone app is available for smartphones running on the Android and iOS operating systems and it is installed on the personal smartphone of the patient.
* Commercial smart wristband. This is a commercial activity tracking device that will be employed for monitoring the physical activity and the sleep quality of the patient, provided by the site personnel. Wearable to be worn. Ionic™ (Fitbit) will be employed by the trial as the smart wristband.
* MyPal web application (app). This is the main interface of the HCP to the system. It is accessible as a web portal through any modern web browser.
* System backend. This module resides at the backend of the system and it is not directly accessible by the aforementioned types of users. The system backend interfaces the MyPal smartphone app and the MyPal web app.

In brief, the intervention revolves around the reporting by the patient of physical and psycho-emotional symptoms (via the MyPal smartphone app) and the immediate delivery of the reported symptom-related information to the HCP (via the MyPal web app). Of note, the reported symptom-related information becomes instantly available to the HCP in the MyPal web app; however, this does not imply that the HCP is guaranteed to review it at the same time. The intervention is described in more detailed below, first from the standpoint of the patient and then from that of the HCP.

The patients interact with the MyPal smartphone app in 3 sequential phases. Additionally, during the enrollment in the study, the patients are handed the commercial smart wristband and they are instructed to wear it as much as possible (also while sleeping) throughout their participation in the study.

Registration Phase. This phase is completed the first time the patient uses the MyPal smartphone app, which take place right after the patient is enrolled in the study. The mission of this phase is (1) to register the patient into the MyPal system, (2) to initially set a number of preferences, (3) to collect via self-reporting the baseline assessment of the patient's physical and psycho-emotional symptom, and (4) to screen for motivational targets and non-adherence risk. The smartphone app guides the patient throughout the entire registration process in a wizard-like fashion, where the user has to provide some information (1)-(2) and complete certain questionnaires (3)-(4). The latter is elaborated in the next phase.

Main usage phase. As soon as the registration phase is completed, the MyPal smartphone app enters into its main usage phase. This lasts 6 months (Month 0 to Month 6 of the patient's participation in the study) and, during this time, the patient is given access to a number of user-initiated functionalities (i.e., functionalities that the user has access to at all times) and system-initiated ones (i.e., functionalities for which the system decides when they become available to the user). More specifically, the functionalities of the second category are initiated via notifications that are presented by the smartphone app to the user. We can distinguish two main types of notifications, namely the intervention notifications (i.e., notifications associated with functionalities that are part of the interventions) and the assessment notifications (i.e., notifications informing the patient it's time to complete the assessment questionnaires that have been foreseen by the study protocol). The intervention notification frequency is once every a multiple of 1 week (e.g., 1 week, 2 weeks, 6 weeks), depending on the specific system-initiated functionality, while the intervention notifications are issued once per month. Whenever possible, messages concerning multiple functionalities are grouped in a single notification, either intervention notification or mixed one.

Follow-up usage phase. The follow-up usage phase starts immediately after the completion of the main usage phase and it also last 6 months (Month 7 to Month 12 of the patient's participation). This phase is identical to the previous phase (all the previously described functionalities are available) with a single exception. This is that the smartphone app does not issue assessment notification monthly; instead it issues only one such notification at the end of Month 12.

In contrast to the case of the patients, the HCP interact with the MyPal web app (i.e., their interface to the MyPal system) in the same manner throughout their participation in the study (this is considered to be from the first to the last month of the study). The only exception to this (main usage) is a short procedure that registers them into the MyPal system; the registration takes place the first time the HCP accesses the MyPal web app.

In brief, during the main usage of the MyPal web app, the HCP get access to the data that are collected by (1) the MyPal smartphone app and (2) the commercial smart wristband and stored in the system backend. The collected data become available to the MyPal web app as soon as they are stored. At individual level, the HCP is authorized to access only the data of the patients of the associated clinical center; however, access to aggregated and summarized data coming from all the patients (descriptive statistics such as min, max, average and percentiles) will also be provided to all the HCP. In contrast to the notification-heavy approach that was adopted for the patients, the HCP are not actively notified by the MyPal system at any point. To compensate for this, the study protocol mandates that the individual data of the participating patients of a given clinical center are reviewed by the associated HCP at least once every 72 hours. The data review and any action related to this will be recorded through the web interface. The absence of notifications means that all functionalities offered to the HCP are user-initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years)
2. Diagnosed with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) or myelodysplastic syndrome (MDS)
3. Scheduled to receive any line of treatment for CLL/SLL or MDS or who have been previously exposed to any treatment for CLL or MDS
4. Able to understand and communicate in the respective language
5. Users of an Internet connected device (smart phone/tablet)

Exclusion Criteria:

1. Patients who are already participating in another experimental study
2. Patients needing immediate referral for specialized palliative care
3. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
4. Patients unable to provide written informed consent
5. Life expectancy <3 months
6. For CLL cohort: patients who have experienced Richter transformation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in EORTC Quality of Life Questionnaire (QLQ)-C30 General Questionnaire | through study completion, an average of 1 year
  The primary objective is to determine whether - compared to standard care - the MyPal-ADULT intervention can lead to improved QoL as evidenced by statistically significant higher scores in EORTC Quality of Life Questionnaire (QLQ)-C30 General Questionnaire
Improvement in EuroQol (EQ)-five dimensions (5D) | through study completion, an average of 1 year
  The primary objective is to determine whether - compared to standard care - the MyPal-ADULT intervention can lead to improved QoL as evidenced by statistically significant higher scores in EuroQol (EQ)-five dimensions (5D).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Ghia, MD,PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chatzikonstantinou T, Vasilopoulou M, Kyrou D, Karakatsoulis G, Argyropaidas P, Besikli-Dimou S, Bonotis P, Chatzimina M, Didi J, Dimosthenous C, Garani-Papadatos T, Hoffman S, Kakalou C, Kazantzaki E, Kiefer S, Koumakis L, Ling J, Maramis C, Meyerheim M, Payne C, Papangelou C, Payne S, Pontikoglou C, Reston R, Ryblom H, Sander A, Schera F, Smedby KE, Zacharioudakis G, Chatzidimitriou A, Doubek M, Stavroyianni N, Ghia P, Papadaki HA, Rosenquist R, Graf N, Natsiavas P, Stamatopoulos K, Karamanidou C, Scarfo L. Assessing an eHealth Intervention on Quality of Life in Patients With Chronic Lymphocytic Leukemia and Myelodysplastic Syndromes: The MyPal Randomized Controlled Trial. JCO Oncol Pract. 2025 Aug 25:OP2500087. doi: 10.1200/OP-25-00087. Online ahead of print. PMID 40854168
- [Derived] Payne S, Begovic D, Salifu Y, Nelson A, Payne C, Downing J, Natsiavas P, Ling J. Applying Digital Health in Cancer and Palliative Care in Europe: Policy Recommendations from an International Expert Workshop (MyPal Project). J Palliat Med. 2024 Feb;27(2):216-223. doi: 10.1089/jpm.2023.0309. Epub 2023 Sep 22. PMID 37738323
- [Derived] Scarfo L, Karamanidou C, Doubek M, Garani-Papadatos T, Didi J, Pontikoglou C, Ling J, Payne C, Papadaki HAlpha, Rosenquist R, Stavroyianni N, Payne S, Ghia P, Natsiavas P, Maramis C, Stamatopoulos K. MyPal ADULT study protocol: a randomised clinical trial of the MyPal ePRO-based early palliative care system in adult patients with haematological malignancies. BMJ Open. 2021 Nov 2;11(11):e050256. doi: 10.1136/bmjopen-2021-050256. PMID 34728446